CLINICAL TRIAL: NCT04288518
Title: SPECT Imaging of Brain Tumors Using Technetium-99m Labeled 1-Thio-D-Glucose (99mTc-1-thio-D-glucose).
Brief Title: Molecular Imaging of Brain Tumors Using Labeled Technetium-99m 1-Thio-D-Glucose.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Imaging of brain tumors
Record Dates: First submitted 2020-02-19; First posted 2020-02-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Brain; Neoplasms
Keywords: 99mTc-1-thio-D-glucose; Brain; Neoplasms; SPECT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary Brain Tumor (Experimental): The tested injected doses of 99mTc-1-thio-D-glucose 500 megabecquerels (MBq).
  At least five (5) evaluable subjects with primary brain tumor. The tested injected dose 500 MBq.
  Interventions: Drug: SPECT or SPECT-CT with 99mTc-1-thio-D-glucose
- Recurrence of Brain Tumor (Experimental): The tested injected doses of 99mTc-1-thio-D-glucose 500 MBq.
  At least five (5) evaluable subjects with recurrence of brain tumor. The tested injected dose 500 MBq
  Interventions: Drug: SPECT or SPECT-CT with 99mTc-1-thio-D-glucose
- Benign intracranial lesions (Experimental): The tested injected doses of 99mTc-1-thio-D-glucose 500 MBq.
  At least five (5) evaluable subjects with benign intracranial lesions. The tested injected dose 500 MBq
  Interventions: Drug: SPECT or SPECT-CT with 99mTc-1-thio-D-glucose

INTERVENTIONS:
Drug: SPECT or SPECT-CT with 99mTc-1-thio-D-glucose — One single intravenous injection of 99mTc-1-thio-D-glucose, followed by gamma camera imaging directly postinjection and after 2, 4, 6 and 24 hours.
  Other Names: 99mTc-1-thio-D-glucose

SUMMARY:
The study should evaluate the biological distribution of 99mTc-1-thio-D-glucose in patients with primary brain tumors and recurrence of brain tumors.

The primary objective are:

1. To assess the distribution of 99mTc-1-thio-D-glucose in normal tissues and tumors at different time intervals.
2. To evaluate dosimetry of 99mTc-1-thio-D-glucose.
3. To study the safety and tolerability of the drug 99mTc-1-thio-D-glucose after a single injection in a diagnostic dosage.

The secondary objective are:

1. To compare the obtained SPECT imaging results of brain tumors with the data of magnetic resonance imaging (MRI) and/or positron emission tomography (PET) and immunohistochemical (IHC) studies of postoperative material.

DETAILED DESCRIPTION:
The overall goal is to study the effectiveness of SPECT imaging of primary brain tumors and relapse of brain tumors using technetium-99m labeled glucose.

Phase I of the study:

Biodistribution of 99mTc-1-thio-D-glucose in patients with primary brain tumors and in patients with recurrence of a brain tumor.

The main objectives of the study:

1. To evaluate the distribution of 99mTc-1-thio-D-glucose in normal tissues and tumors in patients with brain tumors at different time intervals.
2. To evaluate dosimetry 99mTc-1-thio-D-glucose based on the pharmacokinetic parameters of the drug after a single intravenous administration.
3. To study the safety of use and tolerability of the drug 99mTc-1-thio-D-glucose after a single intravenous administration in a diagnostic dosage.

Additional research tasks:

1. To conduct a comparative analysis of the diagnostic information obtained in the visualization of brain tumors by SPECT using 99mTc-1-thio-D-glucose with data obtained by magnetic resonance imaging (MRI) and/or positron emission tomography (PET) and immunohistochemical (IHC) research of postoperative material.
2. To study the diagnostic effectiveness of 99mTc-1-thio-D-glucose SPECT in imaging of brain tumors.
3. To evaluate the overall survival of patients with brain tumors depending on the results of 99mTc-1-thio-D-glucose SPECT.

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labelled tracer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of a primary brain tumor or recurrence of a brain tumor with immunohistological verification.
* Clinical and radiological diagnosis of a benign intracranial lesions.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* alanine amino transferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST): =< 5.0 times Upper Limit of Normal
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Second, non-brain malignancy
* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
* Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body 99mTc-1-thio-D-glucose uptake value (percent) | 24 hours
  Whole-body 99mTc-1-thio-D-glucose uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (percent) of the injected dose of the radiopharmaceutical
SPECT-based 99mTc-1-thio-D-glucose value in tumor lesions (counts) | 6 hours
  99mTc-1-thio-D-glucose uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based 99mTc-1-thio-D-glucose uptake value (counts) | 6 hours
  Focal uptake of 99mTc-1-thio-D-glucose in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (unitless value) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-1-thio-D-glucose uptake coinciding with tumor lesions (counts) will be divided by the value of 99mTc-1-thio-D-glucose uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Safety attributable to 99mTc-1-thio-D-glucose injections, based on the rate of abnormal physical findings (percent) | 24 hours
  The safety attributable to 99mTc-1-thio-D-glucose injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (percent of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-1-thio-D-glucose injections, based on the rate of abnormal laboratory results (percent) | 24 hours
  The safety attributable to 99mTc-1-thio-D-glucose injections will be evaluated based on the blood and urine laboratory tests (percent of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-1-thio-D-glucose injections, based on the rate of adverse events (percent) | 24 hours
  The safety attributable to 99mTc-1-thio-D-glucose injections will be evaluated based on the rate of adverse events (percent)
Safety attributable to 99mTc-1-thio-D-glucose injections, based on the need for concomitant medication (percent) | 24 hours
  The safety attributable to 99mTc-1-thio-D-glucose injections will be evaluated based on the rate of administration of concomitant medication (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimr I Chernov, Principal Investigator — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.